CLINICAL TRIAL: NCT03565965
Title: Mental Practice Combined With Physical Practice to Improve the Gait Performance of People With Parkinson's Disease: A Multicentre Randomized Controlled Trial Protocol
Brief Title: Protocol: Mental Practice Combined With Physical Practice of Gait in Parkinson's Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Brasilia (Other); Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pikel 02
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease
Keywords: Randomized clinical trial; Parkinson's disease; Gait disorders; Locomotor imagery training
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): The Experimental training (ET) consists of 10 sessions with 4 blocks of MP (GMP) intercalated with 4 blocks of gait physical practice (GPP), under single (ST) and dual-task (DT) conditions.
  Interventions: Behavioral: Experimental training
- Control Group (CG) (Active Comparator): The Control training (CT) consists of 10 sessions with 4 blocks of MP (nGMP) intercalated with 4 blocks of gait physical practice (GPP), under single (ST) and dual-task (DT) conditions.
  Interventions: Behavioral: Control training

INTERVENTIONS:
Behavioral: Experimental training — Each block of MP consists of 5 mental walking attempts with 10 imagined steps. Participants, seated comfortably, eyes closed, will be asked to imagine themselves walking as of a first-person perspective, without any overt physical movement, in four different conditions: habitual speed, as fast as possible, overcoming obstacles and memorizing a name of a specific medication.
  Each block of PP consists of 5 physical walking attempts, with 10 steps. Participants will be asked to walk in 4 different conditions: habitual speed,as fast as possible, overcoming obstacles and memorizing a name of a specific medication.
  Arms: Experimental Group (EG)
Behavioral: Control training — Each block of MP consists of 5 mental walking attempts with 10 imagined steps. Participants, seated comfortably, eyes closed, will be asked to imagine themselves seated appreciating a beautiful landscape as of a first-person perspective, without any overt physical movement, in four different contexts: in a carriage, in a hot air balloon, in a boat and in a zepelin.
  Each block of PP consists of 5 physical walking attempts, with 10 steps. Participants will be asked to walk in 4 different conditions: habitual speed,as fast as possible, overcoming obstacles and memorizing a name of a specific medication.
  Arms: Control Group (CG)

SUMMARY:
Among the impairments associated with Parkinson's disease (PD), gait disturbance is one of the most injurious to the independence in daily living activities and the quality of life of people living with Parkinson's disease (PPD). Despite a considerable amount of research, there is no consensus about the most efficient physiotherapeutic approach to improve gait disturbance. Mental practice (MP) is considered an efficient strategy to improve the motor performance of healthy individuals and people with stroke. However, there is little evidence about its therapeutic results as a tool to improve gait performance in PPD. Thus, the aim of this study is to investigate the effects of mental gait practice associated with physical practice (PP) to improve the gait performance of PPD.

DETAILED DESCRIPTION:
Background: Among the impairments associated with Parkinson's disease (PD), gait disturbance is one of the most injurious to the independence in daily living activities and the quality of life of people living with Parkinson's disease (PPD). Despite a considerable amount of research, there is no consensus about the most efficient physiotherapeutic approach to improve gait disturbance. Mental practice (MP) is considered an efficient strategy to improve the motor performance of healthy individuals and people with stroke. However, there is little evidence about its therapeutic results as a tool to improve gait performance in PPD.

Objectives: To investigate the effects of mental gait practice associated with physical practice to improve the gait performance of people living with Parkinson's Disease.

Design: Parallel, prospective, double-blind, multicentre randomized clinical trial.

Setting: Brazilian Parkinson Association.

Participants: Onde hundred and forty four people living with Parkinson's disease in stages 2-3 disease evolution according to Hoehn and Yahr Classification.

Interventions: The participants will be randomly allocated in an experimental group (EG), and a control group (CG). Both groups will perform 10 individual training sessions, two individual sessions per week, for five weeks. Every session will be guided by a physiotherapist. The training sessions consist of four blocks of MP intercalated with four blocks of PP of gait in single-task (ST) and dual-task (DT) conditions. The only difference between the groups will be the content of mental practice blocks: the EG will perform mental practice of gait (GMP) while the CG will perform non-gait mental practice (nGMP).

Randomization: Participants will be randomized by ClinStat software into one of two groups: Experimental Group (EG), which will perform the GMP; and Control Group (CG), which will perform the nGMP.

Statistical analysis: The training effects for each primary and secondary outcome measure will be analyzed for the two training conditions (i.e., control and experimental) at the four assessment time points (i.e., 7 days pre-intervention and post-completion, and at 30 and 60-day follow-up) using a mixed-design ANOVA with training as the between-group factor and the assessment time point as the within-group factor. The effect sizes (ES) will be calculated for all comparisons at alpha = 0.05. A Tukey HSD post-hoc test will be used for multiple comparisons and p-values below 5 % will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's disease according to the United Kingdom Brain Bank criteria;
* in stage 2-3 of the disease evolution according to the Hoehn and Yahr;
* treated with levodopa or its synergists;
* capable to walk independently indoors without aid;
* referring 5 years of education or more.

Exclusion Criteria:

* presence of other neurological (excluding PD), orthopedic or cardiopulmonary problems;
* visual and auditory deficiency uncorrected;
* dementia [assessed by Montreal Cognitive Assessment (MoCA), cut-off 26];
* depression [according to the Geriatric Depression Scale (GDS-15), cut-off 6];
* declined imagery capacity [according to the Revised Movement Imagery Questionnaire (MIQ-R) cut-off 10].

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Postural Instability and Gait Difficulty Score | up to 3 months
  The Postural Instability and Gait Difficulty Score (PIGD) is a recommended rating scale for evaluation of gait alterations in PD based on 5 Unified Parkinson's Disease Rating Scale (UPDRS) items relevant to gait and postural instability (items 13-15, 29, and 30). The 13-15 items are based on gait performance according to PPD perspective, while 29 and 30 items are based on the motor test.
Six-minute Walk Test | up to 3 months
  The six-minute walk test (6-MWT) is a timed recommended clinically based test in which participants are asked to walk for 6 minutes, in their habitual speed, as much distance as possible. Interruptions for resting are permitted if necessary. The 6-MWT has demonstrated adequate test-retest and interrater reliability and minimal detectable change of 82 meters in PD. It may be a good predictor of the ability to independently walk outside safely.
Dynamic Gait Index | up to 3 months
  The Dynamic Gait Index (DGI) is a test that assess gait balance. It has demonstrated good feasibility, test-retest, interrater reliability and minimal detectable change of 3-point reduction in PD. Furthermore, it is considerable as a supportive test for identifying the fall risk in people with PD. The balance during the eight gait related activities is scored in this test. These include quality of walking speed change, going around and over obstacles and stair walking, as well as the number of steps required for a pivot turn. The performance is scored from 0 to 3, with 0 indicating the lowest and 24 the highest level of functioning.
30 seconds DT gait | up to 3 months
  The 30 seconds DT gait (30sDTG) is a test in which measures the maximal walking distance reached in 30 seconds under single and dual taks. The cognitive task consists of speaking as many words as possible, starting with a specific character (F, S or A), presented at the beginning of test. This cognitive task showed to be more sensitive for dual task impairment and less prone to education level.
Functional Near Infrared Spectroscopy (fNIS) | up tp 3 months
  During 30sDTG, the concentration of oxygenated and deoxygenated hemoglobin of the motor and prefrontal regions will be measured. The measuring cap based on the 10-20 international will be set to acquire signal from primary motor cortices and dorsolateral prefrontal cortices. Data will be modelled based on the onset gait time for 30s, automatically defined by trigger markers. The onset and duration of each condition will be convolved with the canonical hemodynamic response function to obtain the regressors. The individual and group measures comparisons, considering the condition with and without dual task will be performed with a significance level of 5%.

SECONDARY OUTCOMES:
Trail Making Test | up to 3 months
  The Trail Making Test (TMT) is s a well-established test constituted for two timed parts: Part A, which involves a visual-scanning task where the participant is required to draw lines sequentially connecting consecutively numbered circles (1-25) randomly arranged on a page as fast as possible. Part B, which measures of cognitive flexibility, where the participant is asked to connect the same number of circles in an alternating sequence of numbers and letters (1, A, 2, B, etc.). In order to avoid the effect of motor speed on the test performance, the time difference between parts (Part B - Part A) is usually used as the more accurate measure of executive function than the performance in one of the parts alone. The time difference between Part B and Part A has showed high correlation with obstacle course gait speed, and with the ability to appropriately adapt gait to environmental challenges in older individuals, and with poor balance and gait performance in PPD.
39-item Parkinson's Disease Questionnaire | up to 3 months
  The 39-item Parkinson's Disease Questionnaire (PDQ 39) is a scale that assesses the health-related quality of life. It evaluates 39 parameters in eight groups of issues (mobility, daily living activities, emotional well-being, stigma of the disease, back in the next, cognitive, communication and bodily discomfort). Each group is constituted from 3 to 10 parameters with five possible answers.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisa P Piemonte, PhD, Principal Investigator — Department of Physioterapy , Communication Science&Disorders, Occupational Therapy, School of Medicine, University of São Paulo
Locations (1):
- Brazil Parkinson Association, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided